CLINICAL TRIAL: NCT01183546
Title: Biomechanical Validation of the Transfer Assessment Instrument (TAI)
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: B7149-I
Record Dates: First submitted 2010-07-16; First posted 2010-08-17 (Estimated); Results first posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-02

CONDITIONS: Spinal Cord Injury
Keywords: rehabilitation; spinal cord injury; wheelchairs
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Wheelchair Users with Spinal Cord Injury: wheelchair users with spinal cord injury

SUMMARY:
The purpose of this research study is to further develop and refine the Transfer Assessment Instrument (TAI). The TAI is a clinical tool to be used by therapists to evaluate transfer techniques and performance.

DETAILED DESCRIPTION:
For Veterans who rely on wheelchairs for mobility, performing transfers is essential to achieving independence with activities of daily living. For example, transfers are required for getting into and out of bed, on and off a bath tub/shower seat, commode seat, motor vehicle seat and so on. Unfortunately transfers, along with wheelchair propulsion, weight relief and overhead activities are believed to largely contribute to the development of shoulder pain and injury. For individuals who rely are their arms for independence with ADL, the onset of pain or an overuse injury can be devastating leading to increased healthcare expenses, limitation in activity, depression, decreased societal participation and a reduced quality of life. Despite the importance of transfers to daily living and that transfers rank among the most strenuous wheelchair-related activities, there is a paucity of research on the biomechanics of transfers.

During rehabilitation, achieving transfers in the safest and most efficient manner possible has traditionally been the goal of both the patient and clinician. However, there is wide variation in the amount and quality of transfer training that is provided in rehab. The ergonomics of performing transfers is crucial to maintaining maximal upper limb function and pain free limbs over time. The techniques taught to patients during rehab are not based on scientific evidence and there is not a uniform way of measuring performance. For these reasons, the investigators developed the Transfer Assessment Instrument (TAI) a 29-item criterion-referenced construct comprised of three domains 1) preparing for a transfer, 2) use of conservation techniques, and 3) quality of the transfer. The instrument was designed to be used by therapists in the clinic to determine a patient's adherence with 'best' transfer techniques, identify targeted areas of intervention, and document performance outcomes pre-post transfer training, intervention (e.g. trunk orthosis) or change in medical status. The TAI includes items that address the ergonomics of transferring independently and dependently for patients who need assistance either from a caregiver or with transfer equipment.

The intent of the proposed three-year study is to establish the psychometric rigor of the TAI with wheelchair users with SCI using a two-phase approach. In Phase 1, 100 subjects will be evaluated for initial psychometric analysis and tool refinement. In Phase 2, using the refined tool extensive biomechanical validation studies will be conducted with 70 individuals who independently perform wheelchair transfers. Tool validation is an important first step towards the effective translation of evidence-based practices into a clinical setting. As a result, the proposed work has great potential to improve the quality of care of veteran patients and reduce the incidence of upper limb pain and injuries.

ELIGIBILITY:
Inclusion Criteria:

For preliminary phase (control subjects)

1. 18 years old or over
2. Ability to do a seated push up (from a seated position, elevate torso and lift buttocks off of the seat using the upper limbs)

For final phase (case subjects)

1. 18 years old or over
2. C4 level or below spinal cord injury
3. Ability to perform an independent transfer (without assistive device or human assistance)
4. Manual wheelchair user For preliminary phase (control subjects)

(1) No significant upper extremity pain or injury that would inhibit the ability to perform transfers or weight bear on the upper extremities.

Exclusion Criteria:

For final phase (case subjects)

1. No significant upper extremity pain or injury that would inhibit the ability to perform transfers or weight bear on the upper extremities.
2. A history of cardiopulmonary (heart/lung condition) that may be exacerbated.
3. Active pressure sores, or a history of pressures sores that may be exacerbated.
4. Functional motor control in the lower extremities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: To initially evaluate the transfer measurement system and protocol, individuals without disability will be recruited (preliminary phase). After validating and evaluating the reliability and sensitivity of the measurement system, individuals with paraplegia and tetraplegia will be recruited (final phase).
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alicia M Koontz, PhD, Principal Investigator — VA Pittsburgh Health Care System
Locations (1):
- VA Pittsburgh Health Care System, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Wheelchair Users With Spinal Cord Injury
Started | 53
Completed | 53
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Wheelchair Users With ASIA A or B Spinal Cord Injury: wheelchair users with ASIA A or B spinal cord injury
Arm/Group | Wheelchair Users With ASIA A or B Spinal Cord Injury
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 53
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 40
Region of Enrollment [Number; unit: participants]
  United States | 53

OUTCOME MEASURES:

1. Primary Outcome: Transfer Performance (TAI Scores Part 1)
Description: Part 1 of the TAI is comprised of 15 items which are scored "yes" (1 point) when the subject performs the specified skill correctly and "no" (0 points) when the subject performs the skill incorrectly or "(N/A)" which means the item does not apply. The part 1 summary score is the summation of each item's score multiplied by 10, and then divided by the number of applicable items, ranging from 0 to 10.
Time Frame: Baseline Testing and at Followup Testing (4 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline Transfer Testing: Wheelchair Users with Spinal Cord Injury who met criteria for transfer training
- Followup Transfer Testing: Wheelchair users with spinal cord injury who met the criteria for transfer training at Baseline and returned four weeks later for transfer training and retesting.
Arm/Group | Baseline Transfer Testing | Followup Transfer Testing
Number analyzed (Participants) | 11 | 11
units on a scale | 6.31 (0.98) | 9.92 (0.25)

2. Secondary Outcome: Shoulder Peak Resultant Moment
Description: Shoulder Peak Resultant Moment during wheelchair transfers was calculated using an inverse dynamics model approach. Inputs into the model included forces recorded at the hands during transfers, three-dimensional motion trajectories of markers placed on the upper limbs and trunk, and subject's anthropometric data.
Time Frame: Baseline Testing and at Followup Testing (4 weeks)
Measure: Mean (Standard Deviation); unit: Newton-meter/kilogram
Arm/Group | Baseline Transfer Testing | Followup Transfer Testing
Number analyzed (Participants) | 11 | 11
Newton-meter/kilogram | 0.97 (0.35) | 0.62 (0.23)

ADVERSE EVENTS:
Arm/Group | Wheelchair Users With ASIA A or B Spinal Cord Injury
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No